CLINICAL TRIAL: NCT06482957
Title: CAUSAL: Cohort to Augment the Understanding of Sarcoma Survivorship Across the Lifespan
Brief Title: Cohort to Augment the Understanding of Sarcoma Survivorship Across the Lifespan
Acronym: CAUSAL
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Debra Friedman, Professor of Pediatrics (Pediatric Hematology and Oncology), Vanderbilt-Ingram Cancer Center
Other Study IDs: VICCPED2222; NCI-2023-00569 (Registry Identifier: NCI, Clinical Trials Reporting Program); 1UG3CA260318-01 (NIH)
Record Dates: First submitted 2024-06-12; First posted 2024-07-01 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Surveys and Questionnaires; Blood Specimen Collection; Urine Specimen Collection; Tissue Banks

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Patients monitor physical activity, sedentary behavior, heart rate and sleep wearing a FitBit device, undergo blood urine, stool and/or saliva sample collection, complete surveys and have medical records reviewed throughout study.
  Interventions: Other: Surveys; Other: Blood Collection; Other: Saliva Collection; Other: Urine Collection; Other: Stool Collection; Other: Tissue collection; Other: Physical Activity Monitoring

INTERVENTIONS:
Other: Surveys — Complete surveys
Other: Blood Collection — Undergo blood collection
Other: Saliva Collection — Undergo salvia collection
Other: Urine Collection — Undergo urine collection
Other: Stool Collection — Undergo stool collection
Other: Tissue collection — Undergo tissue collection
Other: Physical Activity Monitoring — FitBit will be worn to track physical activity

SUMMARY:
This study evaluates the impact that a sarcoma diagnosis and treatment have had on patients over time.

DETAILED DESCRIPTION:
* To evaluate the incidence and prevalence and the impact of disease, treatment, sociodemographic and lifestyle contributors on adverse oncologic outcomes (lack of response, recurrence) and non- oncologic outcomes (physical and psychosocial function, financial toxicity, short and long-term organ toxicity) and mortality in the cohort.
* To evaluate the role of drug metabolism and DNA repair genes via functional polymorphisms, known toxicity associated polymorphisms and genetically predicted gene expression levels, as well as polygenic risk scores, on treatment efficacy, cancer therapy-induced normal tissue toxicity and mortality.
* To identify genomic drivers of sarcoma and to use this information to develop personalized liquid biopsy assays for monitoring treatment response, recurrence, and minimal residual disease (MRD) and mortality.
* Evaluate family functioning, psychosocial wellbeing, and financial toxicity.

OUTLINE: This is an observational study.

Patients monitor physical activity, sedentary behavior, heart rate and sleep wearing a FitBit device, undergo blood urine, stool and/or saliva sample collection, complete surveys and have medical records reviewed throughout study.

ELIGIBILITY:
Patients at any age with a history of sarcoma, with or without evidence of a persistent disease

• For pediatric patients

* Parent/primary caregiver of patient
* Sibling of patient aged 8 years or older

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients at any age with a history of sarcoma, with or without evidence of a persistent disease and parent/caregiver of pediatric patients and siblings of patients 8 years or older
Sampling Method: Non-Probability Sample
Enrollment: 2100 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Impact of disease on adverse oncologic outcomes | Approximately six years
  Medical record review of Common Terminology Criteria for Adverse Events (CTCAEs)
Impact of treatment on adverse oncologic outcomes | Approximately six years
  Medical record review of Common Terminology Criteria for Adverse Events (CTCAEs)
Impact of sociodemographic contributors on adverse oncologic outcomes | Approximately six years
  Patient-Reported Outcomes Measurement Information System (PROMIS) Scores
Impact of lifestyle contributors on adverse oncologic outcomes | Approximately six years
  Patient-reported outcome

CONTACTS AND LOCATIONS:
Overall Officials: Debra Friedman, MD, Principal Investigator — Vanderbilt University/Ingram Cancer Center
Locations (1):
- Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee, United States